CLINICAL TRIAL: NCT02546466
Title: Effects of Functional Taping Compared to Sham and Minimal Intervention Strategy on Pain Intensity and Static Postural Control in Patients With Non-specific Chronic Low Back Pain: a Protocol for a Randomized Sham-controlled Trial
Brief Title: Effects of Functional Taping on Static Postural Control in Patients With Non-specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thais Cristina Chaves, Professor, Department of Neuroscience and Behavioral Science at the Ribeirão Preto Medical School at the University of Sao Paulo. Coordinator, Laboratory of Interdisciplinary Research on Musculoskeletal Pain., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 045641/2015
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain
Keywords: low back pain; functional taping; balance; posture; rehabilitation; psychosocial factors; minimal intervention strategy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Functional Star-shape taping (FST) (Experimental): For the Functional Star-shape taping (FST) procedure, four tapes will be applied in the form of an elastic ''I'' with the aim of facilitating muscle activation. The taping will be applied when the participant is in a seated position. The taping will be positioned covering the entire lumbar region and lower part of the thoracic region (T11, T12), and placed first at the center and then on the ends (Castro-Sanchez et al. 2012).The tension of the taping was 25%, this protocol being recommended by the Kinesio taping manual to facilitate muscle activation (Castro-Sanchez et al. 2012; Kase et al. 2003). The participant will remain for on week with FT.
  Interventions: Procedure: Functional Star-shape taping (SFT)
- Sham Functional Taping (Sham-FT) (Sham Comparator): For the Sham-FT procedure, a single bandage 20 cm in length was positioned horizontally, passing through the spinous process of the second lumbar vertebra (Castro-Sanchez et al. 2012). The tension of the taping was 25%, this protocol being recommended by the Kinesio taping manual to facilitate muscle activation (Castro-Sanchez et al. 2012; Kase et al. 2003). The participant will remain for on week with FT.
  Interventions: Procedure: Sham Functional Taping (Sham-FT)
- Minimal Intervention Strategy (MIS) (Active Comparator): The MIS group will receive an educational and counseling booklet (The Back Book) as recommend by Dupeyron et al. (2011) containing information about the low back pain clinical features, risk factors and prognosis, fear avoidance beliefs, how to deal with an acute pain crisis, the early resumption of normal or vocational activities, even when still experiencing pain, and the importance of improvement in functional activity levels and posture, not just pain relief (Delitto et al. 2012). Participants from this group will not receive FT intervention and the investigator will encourage participants to not receive any kind of treatment during the one month epoch after the initial assessment. They will be followed by one of the investigators that will make phone calls to clarify doubts and reinforce the counseling.
  Interventions: Behavioral: Minimal Intervention Strategy (MIS)

INTERVENTIONS:
Procedure: Functional Star-shape taping (SFT) — For the SFT procedure, four tapes will be applied in the form of an elastic ''I'' with the aim of facilitating muscle activation. The taping will be applied when the participant is in a seated position. The taping will be positioned covering the entire lumbar region and lower part of the thoracic region (T11, T12), and placed first at the center and then on the ends (Castro-Sanchez et al. 2012).The tension of the taping was 25%, this protocol being recommended by the Kinesio taping manual to facilitate muscle activation (Castro-Sanchez et al. 2012; Kase et al. 2003). The participant will remain for on week with FT.
  Arms: Functional Star-shape taping (FST)
Procedure: Sham Functional Taping (Sham-FT) — For the Sham-FT procedure, a single bandage 20 cm in length was positioned horizontally, passing through the spinous process of the second lumbar vertebra (Castro-Sanchez et al. 2012). The tension of the taping was 25%, this protocol being recommended by the Kinesio taping manual to facilitate muscle activation (Castro-Sanchez et al. 2012; Kase et al. 2003). The participant will remain for on week with FT.
  Arms: Sham Functional Taping (Sham-FT)
Behavioral: Minimal Intervention Strategy (MIS) — The MIS group will receive an educational and counseling booklet (The Back Book) as recommend by Dupeyron et al. (2011) containing information about the low back pain clinical features, risk factors and prognosis, fear avoidance beliefs, how to deal with an acute pain crisis, the early resumption of normal or vocational activities, even when still experiencing pain, and the importance of improvement in functional activity levels and posture, not just pain relief (Delitto et al. 2012). Participants from this group will not receive FT intervention and the investigator will encourage participants to not receive any kind of treatment during the one month epoch after the initial assessment. They will be followed by one of the investigators that will make phone calls to clarify doubts and reinforce the counseling.
  Arms: Minimal Intervention Strategy (MIS)

SUMMARY:
Background: Low back pain is a major public health problem that affects most people at some point in life, and results in major psychosocial, economic, functional and physical consequences that can last for days and months. Most cases are undiagnosed and become chronic non-specific low back pain. Studies showed that these patients presented changes in postural control, yet the information is inconsistent, as well as the effects of Functional Taping (FT).

Objectives: The aim of this study will be to investigate the immediate and one-month follow-up effects of the use of Functional Taping to lumbar spine on pain intensity and postural control in patients with chronic nonspecific low back pain (CLBP).

Methods: This study will be a sham-controlled and randomized clinical trial. Participants: One hundred and twenty participants (18 and 50 years) both genders. Interventions: Participants will be randomly allocated to receive three possible interventions: Functional Star-shape Taping, Sham Functional Taping (both interventions during seven days) and a Minimal Intervention (MI) (one session). Main outcome measures: Primary outcomes will be pain intensity and posturography to assess balance parameters. Low back pain related disability, global perceived effect of treatment and fear avoidance beliefs will be considered as secondary outcomes. Four measurements of static posturography will be conducted: pre-intervention, immediately after application of the tape, after seven days post-intervention (after removal of the tape) and after one month follow-up period. Secondary and primary outcomes will be assessed on three occasions: pre-intervention, seven days post-intervention and after one month follow-up period. All statistical analysis will be conducted following the principles of intention to treat, and the effects of treatment will be calculated using linear mixed models.

DETAILED DESCRIPTION:
BACKGROUND

Considering that evidence suggests that patients with CLBP have changes in postural control, we highlight the importance of conduct studies to identify treatment strategies that can influence postural control like as FT. In this way, the objective of the present study is to compare the effects of Functional Star-shape Taping (FST) vs. Sham-FT vs. MI on pain intensity and postural control (primary outcomes) in CLBP patients. The secondary outcomes will be low back pain related disability, global perceived effect of treatment and fear avoidance beliefs.

METHODS

Study design

This study will be a sham-controlled, randomized, three-arm parallel-group clinical Study participants

The sample will be composed of 120 participants (both genders) with nonspecific CLBP, who will be referred to the physiotherapy clinic of the UENP Center for Health Sciences (Paraná state, Brazil).

Allergy test

Firstly, an assessor blinded to the treatment allocation collected the baseline data and performed an allergy test on all participants. This allergy test consisted of applying a small patch of FT over the skin. Participants kept this patch on for 24 hours and will be instructed to remove the patch and call the researchers if any allergic reaction occurred. Only patients without allergic reaction to the patch test were then scheduled to undergo randomization.

Randomisation and allocation

The proposed study will follow the recommendations described in Consolidated Standards of Reporting Trials (CONSORT) statement (Moher et al., 2010). Once the patient has accepted an invitation to participate, they will give written consent before being assessed for eligibility. Firstly, one researcher will gather the clinical assessment and allergy test to exclude noneligible participants. Only patients without allergic reaction to the patch test will be scheduled to randomisation. After this initial assessment, participants will be randomly assigned following simple randomisation procedures (computerized random numbers) to 1 of 3 treatment groups (opaque sealed envelopes containing cards will be used): (1) Functional Star-shape Taping (FST), (2) Sham-FT and (3) (MI). The allocation sequence will be generated by a researcher not involved in the assessment and interventions, and one research assistant will assign participants to interventions.

Procedures

Following the allocation process, a blinded investigator will conduct clinical assessments and collect primary and secondary outcomes and psychosocial variables. In the same session, another investigator who is a certified Kinesio tape practitioner, will proceed with the treatment according to the group assignment, and will be therefore responsible for applying the functional tape and MI. Patients in the FST and Sham-FT groups will be blinded to interventions (sham or not) and will be advised to leave the tape in situ for one week. The MI group will receive a booklet with biopsychosocial education and orientations.

Initial evaluation

The evaluations will be carried out according to the recommendations of the Initiative on Methods, Measurement and Pain Assessment in Clinical Trials (IMMPACT) for chronic pain.

Primary Outcomes

Pain intensity

Measurement of pain intensity will accomplish using the application of the NPRS, which consists of a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable".

Postural control on force platform - Static Posturography with and without a secondary task

Static posturography will be evaluated using a force platform (400 Biomec, EMG system of Brazil Ltda®, São José dos Campos, Brazil), with frequency acquisition of 100 Hz and a second-order 35 Hz low pass Butterworth filter. Posturography analysis of the COP will be carried out by four main parameters of balance: (1) ellipse (95%) of the COP in square centimeters (A-COP in cm2); (2) Root Mean Square of oscillation of the COP (RMS in cm2); (3) mean speed (MVeloc in cm/s) of the displacement of the COP in anteroposterior (A/P) and medial-lateral (M/L) directions; and (4) mean frequency (MF in Hz) of the displacement of the COP in anteroposterior (A/P) and medial-lateral (M/L) directions.

A modified clinical test of sensory interaction for balance (CTSIBm) will be used by measuring the static balance in four sensory conditions: (1) eyes open on stable surface; (2) eyes closed on stable surface; (3) eyes open on unstable surface; (4) eyes closed on unstable surface. For each condition, the participant will be evaluated three times for 40 seconds with a 30-second interval between assessments.

For the assessment of static posturography with a secondary task, volunteers will be requested to perform a fast movement of shoulder flexion (bilateral). Participants will be trained to carry out the tests with maximum arm speed (approximately 120º/seg) and amplitude at about 60º immediately after the auditory stimulus. Participants will perform five movements (open and closed eyes), with a time interval of 30 seconds between each repetition and an auditory stimulus will precede the trigger by a random period of 0.5-2 s.

Secondary Outcomes

Disability and Participant ratings of global improvement and satisfaction with treatment - Global perceived effect Fear avoidance beliefs questionnaire (FABQ).

Psychosocial Measures - Baseline measure

Hospital anxiety and depression scale - HADS and Pain catastrophizing scale - PCS and Chronic Pain Self-Efficacy Scale - CPSS.

Interventions

Functional Taping Intervention

Participants will be subjected to one of two possible intervention procedures with FT: 1) Functional Star-shape Taping (FST); 2) Sham Functional Taping (Sham-FT). The participants will be blinded as to whether they received SFT, or Sham-FT, and the two interventions will be performed in the lumbar region. The elastic adhesive bandage used will have 5.0 cm wide and 0.5 mm thick (Kinesio Tex Gold® brand, Kinesio Holding Corporation, Albuquerque, USA) and resistant to contact with water. All participants will be informed that they would receive one of the two types of FT application. During this period of application, the participants will be directed to maintain their daily life activities, and will be blinded with respect to which intervention procedure they received (if sham or not).

Minimal Intervention Strategy (MI)

The MI group will receive an educational and counseling booklet (a booklet based on The Back Book).

Data analysis

The two primary outcome variables (posturography and pain intensity) were considered for calculation of sample size. For posturography, we will consider an improvement of at least 20% mean speed of oscillation of the COP pre- and immediate post-treatment. The sample size was 27 participants. The following specifications were considered: α=5% and 95% statistical power and effect size of 0.76 for F-test. For pain intensity, an improvement of at least 20% on the NPRS (pre-treatment: 5.6 and post-treatment and follow-up: 4, SD = 1.8). The sample size obtained was 93 (31 participants per group). The following specifications were considered: α=5% and statistical power of 95% and effect size of 0.41 for F-test. Thus, to ensure a power suitable and assuming sample losses, 120 participants will be considered (at least #9 losses per group) (GPower 3.0.10, University of Kiel, Germany).

The statistician will be given grouped data, but data will be coded so that the statistician will remain blinded to patients' group allocation and to protect patient confidentiality. The mean effects of the interventions and the group differences for all outcomes (primary and secondary) will be calculated using linear mixed models that incorporated terms for the treatment groups, time (post-intervention and follow-up), and interaction terms (treatment subgroups and time) as well as psychosocial variables, sex and age as covariates. Secondary analysis will be conducted using regression models to determine whether baseline scores of psychosocial variables (HADS, PCS, CPSS) will moderate the effect of treatments (FT, sham FT or MI). The analyzes will follow the intention-to-treat principles.

Additionally, analyzes will be performed on subgroups of patients with worse and better postural control parameters by determining cut-off values for instability based on data previously published in the literature. These analyzes will be carried out to identify potential subgroups of better and worse rates of postural control and possible effects of FT. The same procedure will be performed to analyze psychosocial subgroups.

For all of these analyzes, we will use the IBM SPSS software package, version 22 (IBM Corp, Armonk, New York).

ELIGIBILITY:
Inclusion Criteria:

* (1) aged between 18 and 50 years;
* (2) medical diagnosis of chronic non-specific low back pain in the last 3 months and/or pain during at least half of the days in the past 6 months (Deyo et al. 2014), that is located between T12 and the gluteal folds;
* (3) pain intensity equal to or greater than three;
* (4) pain caused by certain postures, activities and movements; and
* (5) score greater than 14% on the Oswestry Lumbar Disability Index (Vibe Fersum et al. 2013).

Exclusion Criteria:

* (1) red flags (neoplastic diseases or tumors in the spine, inflammatory diseases, infections and fractures);
* (2) serious neurological (or central and peripheral neurological) symptoms, psychiatric, rheumatologic and cardiac diseases;
* (3) disc herniation;
* (4) lumbar stenosis;
* (5) spondylolisthesis;
* (6) history of spinal surgeries;
* (7) pregnancy;
* (8) menstrual period;
* (9) underwent physical therapy treatments (less than 6 months before the evaluation period);
* (10) participants with previously diagnosed balance disorders or with disorders that may interfere with balance (vestibular diseases, whiplash injuries, functional ankle instability or report of "giving" way sensation in ankle during the past 6 months); and
* (11) using medications that alter or cause suppression of sensory perception.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | one month
  Measurement of pain intensity was accomplished by means of the application of the Numerical Pain Rating Scale (NPRS), which consists of a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable." The volunteers will rate their pain based on these parameters.
Postural control on force platform - Static Posturography with and without a secondary task | one month
  For evaluation on the force platform, a modified clinical test of sensory interaction for balance (CTSIBm) (Boulgarides et al. 2003) will be used by measuring the static balance in four sensory conditions: (1) eyes open on stable surface; (2) eyes closed on stable surface; (3) eyes open on unstable surface; (4) eyes closed on unstable surface. For each condition, the participant will be evaluated three times for a period of 40 seconds with a 30 second interval between each evaluation (Ruhe et al. 2011). For an unstable surface, a 13 cm-thick cushion with a density of 5kg/m3 will be used Caffaro et al. (2014).
  For the assessment of static posturography with a secondary task, participant will be requested to perform fast movement of shoulder flexion (bilateral). Participants will perform five movements (open and closed eyes) (Mok et al. 2011).

SECONDARY OUTCOMES:
Disability | one month
  To assess disability from chronic low back pain, the Oswestry Low Back Disability Index, adapted to Brazilian Portuguese by Vigatto et al. (2007) will be used. This instrument consists of 10 items, each of which has six response options. The first response receives 0 points, and describes the absence or a small amount of low back pain and functional disability, while the sixth response, with five points, describes extreme pain or functional disability. The total score was calculated by summing up the points, the largest possible sum being 50. This result will be transformed into a percentage by multiplying it by two. The highest percentage represented greater disability related to back pain.
Fear avoidance beliefs questionnaire (FABQ) | one month
  The FABQ, adapted for Brazil (Abreu et al. 2008), consists of 16 self- response items, and each item was rated on a seven-point Likert scale from 0 (completely disagree) to 6 (completely agree), subdivided into two subscales: one that addressed the fears and beliefs of individuals in relation to work, (FABQ - Work) and one that addressed their fears and beliefs about physical activities (FABQ - Phys). As in the original version, items 1, 8, 13, 14 and 16 were excluded from the sum of the final score, despite being part of the questionnaire. In addition, the score had to be obtained separately on each of the subscales, the distribution of subscale points being related to the work done, summing items 6, 7, 9, 10, 11, 12 and 15 (total ranging between 0 and 42) and the subscale related to physical activities, summing items 2, 3, 4 and 5 (total ranging between 0 and 24).
Participant ratings of global improvement and satisfaction with treatment - Patient Global Impression of Change (PGIC) | one month
  The Patient Global Impression of Change scale is recommended for use in chronic pain clinical trials as a core outcome measure of global improvement with treatment. This measure is a single-item rating by participants of their improvement with treatment during a clinical trial on a 7-point scale that ranges from very much improved to much worse with no change as the mid-point (Dworkin et a. 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrício J Jassi, PhD student, Principal Investigator — Universidade Estadual do Norte do Paraná
Locations (1):
- Universidade Estadual do Norte do Paraná, Jacarezinho, Paraná, Brazil

REFERENCES:
- [Derived] Jassi FJ, Del Antonio TT, Azevedo BO, Moraes R, George SZ, Chaves TC. Star-Shape Kinesio Taping Is Not Better Than a Minimal Intervention or Sham Kinesio Taping for Pain Intensity and Postural Control in Chronic Low Back Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Jul;102(7):1352-1360.e3. doi: 10.1016/j.apmr.2021.03.007. Epub 2021 Apr 2. PMID 33819489
- [Derived] Jassi FJ, Del Antonio T, Moraes R, George SZ, Chaves TC. Effects of functional taping compared with sham taping and minimal intervention on pain intensity and static postural control for patients with non-specific chronic low back pain: a randomised clinical trial protocol. Physiotherapy. 2017 Jun;103(2):154-159. doi: 10.1016/j.physio.2016.05.008. Epub 2016 Jun 14. PMID 27637736